CLINICAL TRIAL: NCT03896282
Title: Outpatient Total Joint Arthroplasty in Dedicated Daycare Facility vs Standard Patient Ward - a Randomized Controlled Trial
Brief Title: Outpatient Total Joint Arthroplasty in Dedicated Daycare Facility vs Standard Patient Ward
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Kirill Gromov, MD, PhD, Ass. professor, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HVH-SDK141-RCT
Record Dates: First submitted 2019-03-27; First posted 2019-03-29 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Arthropathy of Knee; Arthropathy of Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- daycare facility (Active Comparator): After surgery patient stay at daycare facility for mobilisation and stay until discharge or transfer to standard patient ward if nor discharged by 20.000
  Interventions: Other: Mobilization at a dedicated daycare facility
- standard patient ward (Active Comparator): After surgery patients are transferred to standard patient ward for mobilisation and stay until discharge.
  Interventions: Other: Mobilization at a dedicated daycare facility

INTERVENTIONS:
Other: Mobilization at a dedicated daycare facility — All THA's are performed using a standard posterolateral approach with simple posterior soft-tissue repair. No infiltration anesthesia (LIA) is used in THA's. All TKA's are performed with a standard medial parapatellar approach without the use of tourniquet. Physiotherapy is started as soon as possible after surgery in the dedicated day care facility. Time till first mobilization is recorded as is total time mobilized supervised by a physiotherapist before discharge.
  Patients are discharged if fulfilling the discharge criteria before 8 pm. Number of hours spent in hospital in total is recorded.

SUMMARY:
The purpose of this single center randomized controlled trial (RCT) is to investigate whether outpatient arthroplasty surgery in a dedicated daycare facility will improve discharge on day of surgery, as opposed to surgery followed by subsequent stay in the ward and also same day discharge, without compromizing safety and outcome.

DETAILED DESCRIPTION:
Introduction of fast-track total hip arthroplasty (THA) and total knee arthroplasty (TKA) has led to a decrease in length of stay without compromising patient safety and clinical outcome . In recent years outpatient THA and TKA has gained popularity, especially as major focus is placed on reducing cost and increasing efficiency in all medical treatments . Studies have shown outpatient arthroplasty to be feasible both for THA and TKA patients , with up to 70% of unselected patients being potentially eligible for outpatient surgery. Various results are published on success rate of discharged patients on the day of surgery, ranging from 25% to 99% , depending on patient selection and logistic setup. While the majority of published studies utilizes a modern fast-track setup with early mobilization and multimodal pain treatment, the optimal logistic setup remains unknown.

The purpose of this single center randomized controlled trial (RCT) is to investigate whether outpatient arthroplasty surgery in a dedicated daycare facility will improve discharge on day of surgery, as opposed to surgery followed by subsequent stay in the ward and also same day discharge, without compromizing safety and outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical and radiological osteoarthritis of the hip suitable for primary cementless THA and patients with clinical and radiological osteoarthritis of the knee suitable for primary Cruciate Retaining (CR) TKA
* Age 18-80
* American Society of Anesthesiologists (ASA) Score (1-2)
* BMI <35
* Interested in and motivated for same day discharge
* Family or relatives to be present for >24 hours after discharge
* Able to understand and give consent to the study

Exclusion Criteria:

* Unable to provide care at own home on day of surgery for >24 hours after discharge

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Patients discharged on day of surgery | 12 hours
  Success rate of discharge on day of surgery

SECONDARY OUTCOMES:
Patient reported outcomes | 3 months
  Total Oxford hip score (0-48, with 0 being worst and 48 best)
Readmissions | 3 months
  Readmissions within 90 days
Patient reported outcomes | 3 months
  Total Oxford knee score (0-48, with 0 being worst and 48 best)
reoperations | 3 months
  reoperations within 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of Orthopaedic Surgery, Copenhagen University Hospital Hvidovre, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: Undecided